CLINICAL TRIAL: NCT01710982
Title: A Multicentre, Randomised, Double-blind, Placebo-Controlled Study to Evaluate the Safety of TZP-101 (IV Ulimorelin) Administered Post-Operatively in Patients Who Have Undergone Partial Bowel Resection
Brief Title: Study to Evaluate the Safety of Post-Operative TZP-101 (IV Ulimorelin) After Partial Bowel Resection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Norgine (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NPJ5004-04/2011 (SDS)
Record Dates: First submitted 2012-09-14; First posted 2012-10-19 (Estimated); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Postoperative Ileus
MeSH Terms: interventions — ulimorelin; Water; Injections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- TZP-101 (Active Comparator): TZP-101
  Interventions: Drug: TZP-101
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: TZP-101
  Other Names: Ulimorelin HCl monohydrate (ulimorelin·HCl·H2O)
  Arms: TZP-101
Other: Placebo
  Other Names: Placebo (5% dextrose solution in Water for Injection)
  Arms: Placebo

SUMMARY:
A study to evaluate the safety of TZP-101 in comparison with placebo when administered post-operatively in patients who have undergone partial bowel resection.

DETAILED DESCRIPTION:
This was a multicenter, multinational, randomized, parallel, double-blind, placebo-controlled study to evaluate the safety of TZP-101 administered post operatively to male and female patients aged 18-80 years of age who had undergone partial bowel resection.

It was anticipated that 330 patients would be dosed with once-daily IV administration of 480 mcg/kg TZP-101 or placebo on a 2:1 ratio. An approximately 7% loss of eligible patients between randomization and dosing was expected, therefore it was anticipated that approximately 355 patients would be randomized onto the trial.

This study consisted of a screening period, an in-patient treatment period and a follow-up phone call. The follow-up phone call was to be performed 14 days (+/- 2 days) after the last study drug administration and a follow-up clinic visit 32 days after the last study drug administration. The overall study duration for each patient was not expected to exceed 63 days.

Dosing was to be once daily, commencing within one hour following surgery and continuing every 24hrs (+/- 2hrs) until the first BM, up to a maximum of 7 doses for all patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient is 18 to 80 years of age, inclusive.
* Patient is scheduled to undergo open bowel resection.
* Female patients must be postmenopausal (for at least 1 year), surgically sterile, practicing true sexual abstinence, OR must be using adequate contraception (in the opinion of the investigator) for the duration of the study, including the follow-up period (e.g. contraceptive implants, injectables, oral contraceptives, some intrauterine devices [IUD], and/or barrier method (condom or occlusive cap) with spermicidal foam/gel/film/cream/suppository).
* Hormonal and IUD methods of contraception must be established for a period of 3 months prior to dosing and, if changed, alternative methods should be used as directed by the investigator throughout the duration of the study.
* Females of childbearing potential must have a negative pregnancy test at screening and admission

After surgery and prior to administration of the first dose of study drug, the following eligibility criteria must be assessed:

* Patient underwent open bowel resection.
* Patient has given written informed consent

Exclusion Criteria:

* Patient weighs more than 200kg (441 pounds).
* Patient is classified as American Society of Anesthesiologists (ASA) Class 4, 5, or 6
* Patient has complete bowel obstruction.
* Patient is scheduled to receive a low rectal or anal anastomosis (e.g. proctectomy or ileoanal anastomosis) (low rectal is defined as below the anterior peritoneal reflection - typically 9-10cm from the anal verge).
* Patient is scheduled for laparoscopic or laparoscopic hand-assisted procedure.
* Patient's surgical procedure is considered to be an emergency procedure.
* Patient has significant impairment of liver or renal function (alanine aminotransferase (ALT)/ aspartate aminotransferase (AST) 2.5 times the upper limit of normal; creatinine clearance <30mL/minute (min), estimated using serum creatinine with the formula [(140 - age in years) × weight in kg]/[(72 × serum creatinine in mg/dl) × 0.85 for female patients].
* Patient is anticipated to require prolonged post-operative ventilation.
* Patient has a psychiatric disorder or cognitive impairment that, in the opinion of the Investigator, would interfere with participation in the study.
* Patient has participated in an investigational drug study 30 days prior to the study initiation.
* Patient has a positive laboratory test result for controlled substances (other than for those prescribed by a medical professional and/or accounted for by concomitant medications) at screening.
* Patient is known to have Hepatitis B or Hepatitis C infection currently associated with clinically significant symptoms or abnormal liver function.
* Patient has a recent, adult history of clinically significant hypersensitivity reaction(s) to any drug, in the opinion of the Investigator.
* Patient is pregnant (confirmed by pregnancy test) or is breastfeeding.
* Patient has known history of drug or alcohol abuse within the previous year.

After surgery and prior to administration of the first dose of study drug, the following eligibility criteria must be assessed:

* Patient received a low rectal or an anal anastomosis (e.g. proctectomy or ileoanal anastomosis) (low rectal is defined as below the anterior peritoneal reflection - typically 9-10cm from the anal verge).
* Patient underwent a laparoscopic procedure (including a hand-assisted laparoscopic procedure).
* Patient is classified as American Society of Anesthesiologists (ASA) Class 4, 5, or 6.
* Patients has received ulimorelin previously

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2012-02; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Treatment Emergent Adverse Events as a Measure of Safety and Tolerability | 32 days post-dosing
  To evaluate the safety of TZP-101 in comparison with placebo when administered post-operatively in patients who have undergone partial bowel resection.

CONTACTS AND LOCATIONS:
Overall Officials: Sandy Eisen, MD, Study Director — Norgine Ltd